CLINICAL TRIAL: NCT07262814
Title: Efficacy, Safety and Acceptability of Ascending Doses of Arpraziquantel for Opisthorchis Viverrini Infections in Children Aged 2-7 Years: A Single-blind Randomized Placebo-controlled Dose-ranging Trial
Brief Title: Efficacy and Safety of Ascending Doses of Arpraziquantel in Children Infected With Opisthorchis Viverrini
Acronym: ADORA-VI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Lao Tropical and Public Health Institute (Lao TPHI) (Unknown)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADORA-VI
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Opisthorchis Viverrini

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arpraziquantel 30 mg/kg (Experimental): Treatment with a single dose arpraziquantel: 30 mg/kg, orally administered
  Interventions: Drug: Apraziquantel
- Arpraziquantel 40 mg/kg (Experimental): Treatment with a single dose arpraziquantel: 40 mg/kg, orally administered
  Interventions: Drug: Apraziquantel
- Arpraziquantel 50 mg/kg (Experimental): Treatment with a single dose arpraziquantel: 50 mg/kg, orally administered
  Interventions: Drug: Apraziquantel
- Arpraziquantel 60 mg/kg (Experimental): Treatment with a single dose arpraziquantel: 60 mg/kg, orally administered
  Interventions: Drug: Apraziquantel
- Placebo (Placebo Comparator): Placebo treatment, orally administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apraziquantel — Tablets (dispersible) containing 150 mg arpraziquantel
  Arms: Arpraziquantel 30 mg/kg; Arpraziquantel 40 mg/kg; Arpraziquantel 50 mg/kg; Arpraziquantel 60 mg/kg
Drug: Placebo — Tablets containing no active pharmaceutical ingredient (Placebo Tablets)
  Arms: Placebo

SUMMARY:
This study aims to assess the efficacy, safety and acceptability of ascending doses of arpraziquantel compared to placebo in children infected with Opisthorchis viverrini. The primary objective is to determine the dose-response relationship in terms of cure rate. This study will involve children aged 2-7 years, since O. viverrini infections often occur in pre-school and school-aged children, and this group is largely left untreated in current public health programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 7 years (i.e., 24 to 95 months).
* Bodyweight ≥ 10.0 kg
* Written informed consent signed by parents/caregivers (signature or thumbprint).
* Agree to comply with study procedures, including provision of two stool samples at baseline and at follow-up assessment 14-21 days after treatment, respectively.
* Willing to be examined by a study physician prior to treatment.
* At least two slides of the quadruple Kato-Katz thick smears positive for O. viverrini.

Exclusion Criteria:

* Presence or signs of major systemic illness, e.g. severe anaemia (haemoglobin level of < 80 g/L according to WHO) upon initial clinical assessment.
* Known or suspected infection with Taenia solium (cysticercosis).
* Known or suspected acute schistosomiasis.
* Abnormal liver and kidney function.
* Use of anthelminthic drugs within 4 weeks before or during study period.
* Being breastfed.
* Known allergy to study medications (i.e. praziquantel or any of the excipients).
* Being prescribed or taking concomitantly medication with known contraindication or drug interactions with the study medication.
* Concurrent participation in other clinical trials.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate (CR) of arpraziquantel against O. viverrini | 14-21 days after treatment
  CRs will be calculated as the percentage of O. viverrini egg-positive participants at baseline who become egg-negative after treatment.

SECONDARY OUTCOMES:
Egg reduction rates (ERR) of arpraziquantel against O. viverrini | 14-21 days after treatment
  Eggs per gram of stool (EPG) will be assessed by calculating the mean egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of 24. Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs.
Safety and tolerability of the different arpraziquantel dosing regimens, and compared to placebo | 3 hours, 24 hours and 14-21 days after treatment
  Participants will be monitored at the site for 3 hours following treatment for any acute adverse events (AEs). Participants will be interviewed 3 hours and 24 hours after treatment, as well as 14-21days after treatment administration about the occurrence of AEs. AEs will be evaluated descriptively as the difference of proportion reported AEs before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lao Tropical and Public Health Institute (Lao TPHI), Vientiane, Laos